CLINICAL TRIAL: NCT02433392
Title: A Phase 1 Study of Intraparenchymal Therapy With Irinotecan Hydrochloride Drug-eluting Beads (CM-BC2) as an Adjunct Therapy to Best Standard of Care in Patients With Recurrent, Surgically Resectable Glioblastoma Multiforme.
Brief Title: Study of Intraparenchymal Therapy as Adjunct Therapy in Patients With Recurrent, Resectable Glioblastoma Multiforme.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate the trial was based on the slow rate of recruitment across the programme of studies
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA1021
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Glioma
Keywords: drug-eluting beads; irinotecan hydrochloride
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CM-BC2 (Experimental): Patients diagnosed with recurrent, surgically resectable glioblastoma multiforme will receive up to 75 mg irinotecan delivered by drug-eluting beads (CM-BC2).
  Interventions: Procedure: CM-BC2

INTERVENTIONS:
Procedure: CM-BC2 — CM-BC2 is a drug-eluting bead, a drug-device combination

SUMMARY:
The purpose of this trial is to determine the safety and feasibility of injecting irinotecan hydrochloride drug-eluting beads directly into the cavity remaining after a tumor is surgically removed in patients with a type of brain tumor (glioblastoma multiforme - also known as glioma) that has returned after prior therapy.

DETAILED DESCRIPTION:
A challenge in the treatment of glioma is the delivery of treatment to the brain after systemic administration due to the blood brain barrier. To improve drug delivery to the brain to achieve very high local concentrations of the anti-neoplastic agent with low system toxicity, a local regional approach is proposed. CM-BC2, an irinotecan hydrochloride drug-eluting bead, is an investigational medicinal product intended for direction injection into the tumor resection margin. The objective of this trial is demonstration of safety and feasibility of this intraparenchymal injection of irinotecan hydrochloride drug-eluting beads in the treatment of recurrent Glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed diagnosis of Glioblastoma Multiforme (GBM) (World Health Organization grade IV)
2. recurrent disease
3. patient will be considered a good candidate for resection and will have estimated life expectancy of at least 12 weeks as estimated by the Principal Investigator or designee. The decision to opt for resection of the recurrence must be independent of study selection.
4. Tumour characteristics:

   * Single unilateral and supratentorial lesion
   * On clinician's assessment, must be operable under normal considerations of risk vs. benefit for condition and prognosis
5. patient will have received conventional treatment at the time of initial diagnosis, including surgery (biopsy or de-bulking), and/or radiotherapy, and/or chemotherapy
6. male or female; no racial exclusions; at least 18 years of age
7. Pregnancy must be excluded in female patients by beta- HCG (Human Chorionic Gonadotropin); all patients agree to use adequate contraception for study duration
8. Karnofsky Performance Status of at least 60
9. Patients must be able to understand consent and study instructions as well as follow prescribed instructions
10. patient must have signed written informed consent prior to study participation

Exclusion Criteria:

1. patient must not be enrolled in any other clinical trial for 30 days before or after participation in this trial
2. history of allergic reactions attributed to compounds of similar chemical make-up or composition to CM-BC2, alginate or irinotecan; or has any other contraindications to irinotecan therapy
3. open communication between the ventricle CSF (cerebrospinal fluid) and tumour resection cavity/site must be avoided. In the case of opening ventricles during surgery, the surgeon must decide whether effective closure is possible by obstructing the gap with Gelfoam/other appropriate materials
4. Tumor surgery, other than stereotactic biopsy of the GBM, or other neurosurgery within 30 days prior to study entry
5. Multiple GBM lesions
6. Irinotecan chemotherapy within 30 days prior to study treatment
7. radiotherapy or stereotactic (gamma knife) radiosurgery within 90 days prior to study entry
8. loco-regional (intra-cranial) therapy for the treatment of GBM, including administration of biodegradable polymer wafers containing Carmustine and/or brachytherapy, in the 6 months prior to study entry
9. Significant liver function impairment: aminotransferase (AST) or alanine transaminase (ALT) greater than 2.5 x the upper limit of normal (ULN), or total bilirubin greater than 2 x ULN
10. significant renal impairment: creatinine greater than 2.0 mg/dL
11. Coagulopathy Prothrombin time (PT) or partial thromboplastin time (APTT) of less than 1.5 x control, and/or platelet count of less than 100 x 10⁹/L
12. Hb less than 8 g/dL and/or neutrophil count (ANC - Absolute Neutrophil Count) of less than 1 x 10⁹/L
13. Any condition that, in the investigator's opinion, makes it in the patient's best interest not to participate in the study
14. Pre-existing cerebral oedema that, in the surgeon's opinion, poses unacceptable risk of post-operative oedema. This decision may be at time of surgery.
15. Presence of concurrent malignancy, except for adequately controlled limited basal cell carcinoma of the skin or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety measured by incidence of adverse events as assessed by CTCAE v4.0 | 6 months
  safety of intraparenchymal injection of CM-BC2

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  Progression-free Survival (PFS) at 6 months
Systemic serum levels of irinotecan | 6 months
  Serum levels of drug (irinotecan)
Systemic serum levels of SN-38, irinotecan metabolite | 6 months
  Serum levels of drug metabolite (SN-38)

CONTACTS AND LOCATIONS:
Overall Officials: Garth Cruickshank, M.D., Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom